CLINICAL TRIAL: NCT02222662
Title: Phase 1 Study of the Parent-delivered Massage Treatment Protocol for Children With Autism Ages 6 to 11
Brief Title: Parent-delivered Massage for Children With Autism - Ages 6 to 11
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Oregon University (Other)
Collaborators: HRSA/Maternal and Child Health Bureau (U.S. Federal Agency)
Responsible Party: Principal Investigator, Louisa Silva, Principal Investigator, Visiting Professor, Western Oregon University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R40MC24945(2)
Record Dates: First submitted 2014-08-15; First posted 2014-08-21 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2015-12

CONDITIONS: Autism
Keywords: Massage; effectiveness; autism; parent stress
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Parent massage tx group (Experimental): Children in this group receive the parent-delivered massage intervention right after randomization.
  Interventions: Other: Parent massage tx group
- Parent massage wait-list control group (Experimental): Children in this group receive the parent-delivered massage intervention 5 months after randomization.
  Interventions: Other: Parent massage wait-list control group

INTERVENTIONS:
Other: Parent massage tx group — The parent-delivered massage is based on Chinese medicine. There are specific techniques for each area of difficulty, e.g. the head, fingers, and toes. After a few months, massage becomes relaxing and enjoyable, and parent touch comes back into use to effectively help the child self-regulate.
  Arms: Parent massage tx group
Other: Parent massage wait-list control group — The parent-delivered massage is based on Chinese medicine. There are specific techniques for each area of difficulty, e.g. the head, fingers, and toes. After a few months, massage becomes relaxing and enjoyable, and parent touch comes back into use to effectively help the child self-regulate.
  Arms: Parent massage wait-list control group

SUMMARY:
Through funding from the U.S. Maternal and Child Health Bureau, Teaching Research Institute at Western Oregon University (WOU) will be conducting research on the effect of a parent-delivered massage program on measures of autism and general development in children ages 6 to 11 with autism. Families will participate in an initial training, and receive 24 sessions of ongoing support and training from a trained therapist over the first nine months.

DETAILED DESCRIPTION:
Children will be randomly divided into treatment groups and wait-list control groups. The control groups begin treatment five months after the treatment groups begin.

All children will be tested on three occasions in the first year: prior to beginning treatment, and five and twelve months later. Results will be shared with parents at the end of each year. Testers will remain blinded as to which group is currently receiving treatment.

There is no cost to parents for participation in this research study. Families meeting the eligibility criteria will be accepted into the study on a first-come, first-served basis.

ELIGIBILITY:
Inclusion Criteria:

* Have a medical and/or educational diagnosis of autism
* Be between the age of 6 and 11
* Parents willing to attend the parent training session and transport the child to treatment sessions with trained staff 20 times in the first five months
* Parents willing to give the fifteen-minute massage daily
* Parents willing not to start any new interventions unless medically necessary

Exclusion Criteria:

* Taking psychoactive medication or pharmaceutical chelation therapy
* Additional chronic disability (for example, cerebral palsy or uncontrolled seizures)
* Receiving more than fifteen hours per week of intensive behavioral treatment for autism (e.g. Applied Behavior Analysis therapy)

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2014-06; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in severity of autism | 5 months and one year
  The Childhood Autism Rating Scales will be used to measure this.

SECONDARY OUTCOMES:
Change in developmental skills | 5 months and one year
  The Vineland II will be used to measure this.

OTHER OUTCOMES:
Change in communication skills | 5 months and one year
  The Preschool Language Scale-5 will be used to measure this.
Change in co-morbid symptoms of autism | 5 months and one year
  The Sense and Self-Regulation Checklist will be used to measure this.
Change in degree of parenting stress | 5 months and one year
  The Autism Parenting Stress Index will be used to measure this.

CONTACTS AND LOCATIONS:
Overall Officials: Louisa Silva, MD MPH, Principal Investigator — Western Oregon University
Locations (1):
- Various locations in Portland, Salem, Albany/Corvallis and Eugene, Portland, Salem, Albany, Corvallis, Eugene, Oregon, United States

REFERENCES:
- [Background] Silva LM, Schalock M, Ayres R, Bunse C, Budden S. Qigong massage treatment for sensory and self-regulation problems in young children with autism: a randomized controlled trial. Am J Occup Ther. 2009 Jul-Aug;63(4):423-32. doi: 10.5014/ajot.63.4.423. PMID 19708471
- [Background] Silva L, Schalock M. Treatment of tactile impairment in young children with autism: results with qigong massage. Int J Ther Massage Bodywork. 2013 Dec 3;6(4):12-20. doi: 10.3822/ijtmb.v6i4.227. eCollection 2013. PMID 24298297
- [Background] Silva LM, Schalock M, Gabrielsen K. Early intervention for autism with a parent-delivered Qigong massage program: a randomized controlled trial. Am J Occup Ther. 2011 Sep-Oct;65(5):550-9. doi: 10.5014/ajot.2011.000661. PMID 22026323
- [Background] Silva LM, Schalock M, Ayres R. A model and treatment for autism at the convergence of Chinese medicine and Western science: first 130 cases. Chin J Integr Med. 2011 Jun;17(6):421-9. doi: 10.1007/s11655-011-0635-0. Epub 2011 Jun 10. PMID 21660676
- [Background] Silva LM, Schalock M, Gabrielsen KR, Budden SS, Buenrostro M, Horton G. Early Intervention with a Parent-Delivered Massage Protocol Directed at Tactile Abnormalities Decreases Severity of Autism and Improves Child-to-Parent Interactions: A Replication Study. Autism Res Treat. 2015;2015:904585. doi: 10.1155/2015/904585. Epub 2015 Mar 24. PMID 25878901
- See also: Qigong Sensory Treatment Massage for Autism — http://qsti.org